CLINICAL TRIAL: NCT01281098
Title: Prospective, Randomized, Open Label, Phase II Study to Assess Efficacy and Safety of Macugen® (Pegaptanib 0.3 mg Intravitreal Injections) Plus Panretinal Photocoagulation (PRP) and PRP (Monotherapy) in the Treatment of Patients With High Risk Proliferative Diabetic Retinopathy (PDR).
Brief Title: Prospective, Randomized, Open Label, Phase II Study to Assess Efficacy and Safety of Macugen® (Pegaptanib 0.3 mg Intravitreal Injections) Plus Panretinal Photocoagulation and PRP (Monotherapy) in the Treatment With High Risk PDR.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-02-2009; 2009-016760-36 (EudraCT Number)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2013-04

CONDITIONS: High Risk Proliferative Diabetic Retinopathy; Diabetes Mellitus Type I; Diabetes Mellitus Type II
Keywords: High Risk Proliferative Diabetic Retinopathy; Diabetes Mellitus Type I, Type II; Pegaptanib; Panretinal Photocoagulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panretinal Photocoagulation (PRP) (Active Comparator): Group 1: Panretinal photocoagulation treatment (PRP) at week-0 that can be repeated every 6 weeks.
  Interventions: Procedure: Panretinal Photocoagulation (PRP)
- Pegaptanib + Panretinal Photocoagulation (PRP) (Experimental): Group 2: Combination treatment of pegaptanib intravitreous injections at weeks 0, 6 and 12 that can be repeated every 6 weeks. Plus PRP after first injection (2 weeks +/- 1 week)and that can be repeated every 12 weeks.
  Interventions: Procedure: Panretinal Photocoagulation (PRP); Drug: Intravitreous injection of pegaptanib

INTERVENTIONS:
Procedure: Panretinal Photocoagulation (PRP) — Panretinal Photocoagulation (PRP)
Drug: Intravitreous injection of pegaptanib — Intravitreous injection of pegaptanib
  Arms: Pegaptanib + Panretinal Photocoagulation (PRP)

SUMMARY:
To evaluate the safety and determine the efficacy of PRP monotherapy or combination therapy (pegaptanib 0.3 mg plus PRP) in patients with Type I or Type II diabetes mellitus and with high risk proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Panretinal photocoagulation (PRP) can cause regression of retinal neovascularization and reduce the risk of severe vision loss in people with proliferative diabetic retinopathy (PDR). However, this destructive treatment may be associated with side effects (e.g. pain, transient blurring, loss of peripheral and/or night vision, increased risk of macular edema and central vision loss) and it is not always efficient in the regression of the neovascularization.

Vascular endothelial growth factor (VEGF) has been shown to play a role in retinal neovascularization and retinal vascular leakage related with PDR and diabetic macular edema.

Anti-VEGF treatments have been hypothesized as an adjunctive treatment for the management of retinal neovascularization and macular edema related with diabetic retinopathy (DR).

Anti-VEGF agents, such as Macugen®, combined with PRP are expected to control neovascularization without the need for photocoagulation of the posterior pole, around the macula, thus avoiding the major side effects of standard PRP (visual field loss).

A modification of panretinal photocoagulation (PRP) was recently proposed by Madeira et al., (2009) at the 2009 EURETINA Meeting. The described technique involves the progressive application of the DRS photocoagulation rings in a different sequence. First ring: corresponds to the DRS third ring, extruding from the ora serrata to the midperiphery. Second ring: corresponds to DRS second ring, extruding from the midperiphery towards the vortex veins. Third ring: corresponds to DRS first ring, and will only be performed if necessary. This technique resulted in less aggressive visual fields losses by achieving results with only most peripheral photocoagulation. The combination of intravitreal anti-VEGF treatment with pegaptanib, where a series of 3 injections are injected to reverse the neovascularization, while maintaining the macula dry will be completed by the more long term effect of the panretinal photocoagulation. This peripheral photocoagulation proposed is expected to eliminate the chronic VEGF stimulus by eliminating the chronic ischemic factor, while maintaining the visual fields useful for daily activities such as driving, etc.

ELIGIBILITY:
Inclusion Criteria:

* High-risk proliferative diabetic retinopathy (HR-PDR) eyes (as defined in section 2).
* BCVA at baseline > 20/320 (25 letters in the ETDRS Chart) in the study eye.
* Clear ocular media and adequate pupillary dilatation to permit good quality fundus photography.
* Intraocular pressure < 21 mmHg.
* Type I, or Type II diabetic subjects as defined by the WHO criteria of either gender, and aged ≥ 18 years.
* Women must be using effective contraception, be post-menopausal for at least 12 months prior to trial entry, or surgically sterile.
* Ability to provide written informed consent.
* Ability to return for all trial visits.

Exclusion Criteria:

* Eyes with prior scatter (panretinal).
* Focal/grid photocoagulation, within the previous 6 months.
* Fibrovascular proliferation with retinal traction.
* Other cause of retinal neovascularization (retinal vein occlusion, radiation retinopathy or others).
* Atrophy/scarring/fibrosis/ hard exudates involving the center of the macula.
* Subjects who have received YAG laser within the previous 6 months.
* Peripheral retinal cryoablation, or laser retinopexy (for retinal tears only),
* Significant media opacities, which might interfere with visual acuity, assessment of toxicity or fundus photography.
* Subjects should not be entered if there is likelihood that they will require cataract surgery within the following 1 year.
* Any intraocular surgery within 6 months before trial enrolment.
* Previous vitrectomy.
* HbA1C level >11% or recent signs of uncontrolled diabetes.
* Any of the following underlying systemic diseases:
* History or evidence of severe cardiac disease, e.g. NYHA Functional Class III or IV, clinical or medical history of unstable angina, acute coronary syndrome, myocardial infarction, or revascularization procedure within 6 months prior to baseline, or ventricular tachyarrhythmia requiring treatment.

  * History or evidence of clinically significant peripheral vascular disease such as intermittent claudication or prior amputation.
  * Clinically significant impaired renal function (serum creatinine >2.5 mg/dL or s/p renal transplant or receiving dialysis).
  * Clinically significant impaired hepatic function.
  * Stroke (within 12 months of trial entry).
  * Any major surgical procedure within one month before trial enrolment.
* Previous radiation to the head in the region of the study eye.
* Any prior treatment with an investigational agent for diabetic retinopathy or anti-VEGF therapy (including intravitreal, subconjunctival or subtenons corticosteroids) during the past 90 days for any other condition.
* Known serious allergies to fluorescein used in angiography, or to components of Macugen® formulation.
* Systolic BP > 170 (2 different readings) or diastolic BP > 100 (2 different readings).
* Acute ocular or periocular infection.
* Previous filtering surgery (e.g., trabeculectomy) or placement of a glaucoma drainage devise (e.g., tube-shunt surgery).
* Use of other investigational drugs at the time of enrollment.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant UNLESS they are: women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner; women whose partners have been sterilized by vasectomy or other means using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices - IUDs). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) are not acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Regression of retinal neovascularization | 12-month treatment
  Retinal neovascularization will be measured in disc area units, and progression of neovascularization will be defined as an increasing of 0.5 disc area associated or not with vitreous haemorrhage, and/or pre-retinal haemorrhage, and/or rubeosis, and/or traccional retinal detachment.

SECONDARY OUTCOMES:
Changes from baseline in Best-Corrected Visual Acuity (BCVA) | 12-month treatment
  BCVA will be assessed during the trial (Baseline, Month 3,Month 6, Month 12).
Changes from baseline in macular retinal thickness by Optical Coherent Tomography (OCT) | 12-month treatment
  OCT will be assessed during the trial (Baseline, Month 3, Month 6, Month 12).
Changes from baseline in Visual Fields | 12-month treatment
  Visual Fields will be performed during the trial (Baseline, Month 3, Month 6, Month 12).
Recurrence of retinal neovascularization | 12-month treatment
  To assess if there is recurrence of retinal neovascularization.
Number of treatments needed | 12-month treatment
  To analyse the number of treatments given to each subject during the 12-month treatment.
Additional focal or grid laser for DME | 12-month treatment
  To assess the number of subjects that received additional focal or grid laser for DME.
Adverse events | 12-month treatment
  Drug safety profile.
Need for vitrectomy due to occurrence of vitreous hemorrhage or retinal detachment | 12-month treatment
  To assess the number of subjects who needed vitrectomy due to occurrence of vitreous hemorrhage or retinal detachment.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Trials - Aibili, Coimbra, Portugal